CLINICAL TRIAL: NCT06837012
Title: Duloxetine As an Analgesic in Patients Without Central Sensitivity Undergoing Single-sitting, Bilateral Total Knee Arthroplasty: a Prospective, Double-blinded, Randomised, Placebo-controlled Trial
Brief Title: Duloxetine As an Analgesic in Patients Without Central Sensitivity After Same Sitting Bilateral Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Orthopaedic Arthroscopy Knee and Shoulder Clinic (Other)
Collaborators: The Grant Medical College & Sir J.J. Group of Hospitals (Other Government)
Responsible Party: Principal Investigator, Dr. Amyn Rajani, Consultant Orthopaedic surgeon, Department of Orthopaedics, The Grant Medical College & Sir J.J. Group of Hospitals
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MDC/12/12/2020
Record Dates: First submitted 2025-01-28; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis of Knee; Central Sensitization; Central Sensitisation
Keywords: Duloxetine; Total knee arthroplasty; Analgesic; Central sensitisation; Pain; SNRI; Chronic
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Bronchiolitis Obliterans Syndrome | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Duloxetine group (Active Comparator): Patients given duloxetine
  Interventions: Drug: Duloxetine - low dose
- Placebo group (Placebo Comparator): Patients given starch capsules identical in appearance and weight to the duloxetine capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine - low dose — Only patients who underwent single bilateral Total knee arthroplasty and WITHOUT central sensitisation were evaluated
  Arms: Duloxetine group
Drug: Placebo — starch capsules identical in appearance and weight to the duloxetine capsules
  Arms: Placebo group

SUMMARY:
Analgesic effect of 20mg Duloxetine was evaluated at regular short term intervals in patients without central sensitivity and undergoing bilateral single sitting total knee arthroplasty for tricompartmental osteoarthritis using standardised patient related outcome measures like the visual analogue score.

DETAILED DESCRIPTION:
Patients who underwent bilateral, single-sitting total knee arthroplasty for tricompartmental knee osteoarthritis were evaluated preoperatively for having central sensitivity. Only patients without central sensitisation were recruited and randomised into two groups with one group given 20 mg duloxetine capsules and the other group given a starch capsule of same shape, make, and weight as a placebo. Patients were evaluated for pain at rest and movement using VAS. A 6-hourly calculation of VAS was done over the first 48 hours and the average was recorded. Subsequent measurements at 1 week, 2 weeks, 4 weeks, and 3 months after surgery was done by a blinded clinician. Additional, drug safety, NSAID consumption and overall patient satisfaction were studied.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral tricompartmental knee osteoarthritis
* Underwent primary, bilateral TKA in single-sitting

Exclusion Criteria:

* American Society of Anesthesiologists physical status IV
* Hamilton Depression Scale (HAMD) and/or Hamilton Anxiety Scale (HAMA) scores > 7
* known intolerance or allergy to any of the study drugs, alcohol, tobacco, narcotic, or opioid dependence
* patients on anticoagulants
* known hepatic/renal dysfunction
* serious cardiac/cerebrovascular comorbidities
* HbA1c≥7
* patients who were already on duloxetine or other SNRIs, monoamine oxidase inhibitors, tricyclic antidepressants, triptans, lithium, other antiepileptics, or buspirone.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
resting Visual Analogue Score for pain | from enrolment to 3 months after surgery
  The patient has to mark the degree of pain on a scale of 0 to 10 with 10 being the worst pain ever felt and 0 being no pain value were minimum 0 to maximum 10 Higher number denotes more pain and worse outcome
Visual Analogue Score for pain on movement | from enrolment to 3 months after surgery
  The patient has to mark the degree of pain on a scale of 0 to 10 with 10 being the worst pain ever felt and 0 being no pain value were minimum 0 to maximum 10 Higher number denotes more pain and worse outcome

SECONDARY OUTCOMES:
NSAID consumption | from enrolment to 3 months after surgery
  calculated in milligrams of etoricoxib with higher number denoting worse outcome
adverse effects | from enrolment to 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Arthroscopy Knee and shoulder clinic, Mumbai, Maharasthra, India

IPD SHARING:
Plan to Share IPD: No
Can be made available upon reasonable request